CLINICAL TRIAL: NCT01548222
Title: CGM Evaluation of Glucose Excursions in Basal Insulin Treated T2DM at Fasting Glucose Target
Status: Completed | Type: Observational
Sponsor: Diabetes Care Center (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: MM2012
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; continuous glucose; basal insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a trial to determine if patients who are well controlled and on basal insulin are treated with excessive basal dose.

DETAILED DESCRIPTION:
In many clinical trials, basal insulin is titrated to only a fasting glucose goal. The usual final dose is >0.4U/kg. In carefully CGM monitored/titrated studies in both basal insulin alone or in pump-treated T2DM, we have found the basal insulin dose to be <0.3U/kg. This suggests that if guided by a single daily fasting glucose, titration may result in an excessive basal dose. This study will examine that issue.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age 18 years and above
* Concurrently on +/-thiazolidnedione +/-DDP IV inhibitors +/-metformin +/- glinides and basal insulin analogs
* A1C 10% or below
* Capable of self monitoring glucose at least 4 x a day
* Previously compliant with clinical recommendations
* Fasting blood glucose <110mg/dl average for 3 consecutive days
* BMI <45 kg/m

Exclusion Criteria:

* Urinary ketosis
* Current or expected alternation in insulin sensitivity such as major surgery, infection, renal failure, glucocorticoid treatment, recent serious hypoglycaemic episode
* Currently participating in another clinical trial
* Using rapid insulin insulin
* Pregnancy or nursing or the intention of becoming pregnant or not using adequate birth control
* Significant liver or heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the Diabetes Care Center clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of time CGM glucose is <70mg/dl | the subject will be followed for 9 days
  The percentage of time CGM glucose is <70 mg/dl during the basal glucose evaluation

SECONDARY OUTCOMES:
Percentage of time CGM glucose is <40 mg/dl | the subject will be followed for 9 days
  The percentage of time the CGM glucose is <40 mg/dl
Determined hypoglycaemic episodes | the subject will be followed for 9 days
  The percentage of subjects who perceived all CGM determined hypoglycaemic episodes
Weight gain | the subject will be followed for 9 days
  The mean weight gain since initiating basal insulin fromo retrospectively gathered data.

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Care Center, Salinas, California, United States

REFERENCES:
- [Background] Blonde L, Merilainen M, Karwe V, Raskin P; TITRATE Study Group. Patient-directed titration for achieving glycaemic goals using a once-daily basal insulin analogue: an assessment of two different fasting plasma glucose targets - the TITRATE study. Diabetes Obes Metab. 2009 Jun;11(6):623-31. doi: 10.1111/j.1463-1326.2009.01060.x. PMID 19515182
- [Background] Meneghini L, Koenen C, Weng W, Selam JL. The usage of a simplified self-titration dosing guideline (303 Algorithm) for insulin detemir in patients with type 2 diabetes--results of the randomized, controlled PREDICTIVE 303 study. Diabetes Obes Metab. 2007 Nov;9(6):902-13. doi: 10.1111/j.1463-1326.2007.00804.x. PMID 17924873
- [Result] Strange P. Treat-to-target insulin titration algorithms when initiating long or intermediate acting insulin in type 2 diabetes. J Diabetes Sci Technol. 2007 Jul;1(4):540-8. doi: 10.1177/193229680700100412. PMID 19885117
- [Result] King AB. Once-daily insulin detemir is comparable to once-daily insulin glargine in providing glycaemic control over 24 h in patients with type 2 diabetes: a double-blind, randomized, crossover study. Diabetes Obes Metab. 2009 Jan;11(1):69-71. doi: 10.1111/j.1463-1326.2008.01014.x. PMID 19120433